CLINICAL TRIAL: NCT06726291
Title: Akynzeo as Antiemetic Treatment in Patients With Endometrial Cancer Treated With Taxane- Platinum Combination Chemotherapy. NOEME Study.
Brief Title: Akynzeo as Antiemetic Treatment in Patients With Endometrial Cancer
Acronym: NOEME
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INT 121-23 NOEME; 2023-504150-35-00 (EU CTIS Number)
Record Dates: First submitted 2024-11-25; First posted 2024-12-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-11

CONDITIONS: Endometrial Cancer
Keywords: antiemetic; nausea; vomiting; chemotherapy side effects; netupitant/palonosetron
MeSH Terms: conditions — Endometrial Neoplasms; Nausea; Vomiting

STUDY DESIGN:
Intervention Model Description: This is a phase IV, multicentric, single arm study, using a fixed dose combination of netupitant and palonsetron in the treatment of chemo-naive patients ≥18 years of age with histologically or cytologically confirmed diagnosis of endometrial cancer who will receive a single line of taxane-platinum combination with or without immunotherapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- antiemetic (Experimental): Patients who will receive a fixed dose combination of netupitant and palonsetron, NEPA
  Interventions: Drug: NEPA (300mg netupitant/0.5mg palonosetron)

INTERVENTIONS:
Drug: NEPA (300mg netupitant/0.5mg palonosetron) — a single dose (capsule) of NEPA (300mg netupitant/0.5 palonosetron) at day 1 for a maximum of 4 cycles

SUMMARY:
The clinical trial concerns the use of an innovative "anti-emetic" drug (that is, anti-vomiting and nausea) in subjects affected by endometrial cancer. It is addressed to patients who have never received chemotherapy before and are about to start a treatment with platinum and taxanes with or without immunotherapy for endometrial cancer.

The primary objective of the study is to learn if the drug is able to avoid the occurrence of vomiting and post- nausea chemotherapy within 120 hours after cycle 1 with carboplatin and paclitaxel with or without immunotherapy.

Partecipants will take the drug before the chemotherapy/immunotherapy (single dose at day one of each cycle of therapy, that is one capsule before treatment). The entire duration of participation in the study may extend to the fourth cycle of chemotherapy/immunotherapy.

Patients will fill in questionnaires and keep a diary of the number and intensity of symptoms (vomiting and nausea).

DETAILED DESCRIPTION:
Chemotherapy side effects (CSE) have a considerable impact on quality of life and can severely impair a patient's ability to manage daily activities and employment. Moreover, unsatisfactory control of chemotherapy toxicities affecting treatment effectiveness necessitates dose reduction and/or treatment deferral. Measures to reduce CSEs, such as antiemetic drugs and other supportive agents, are often prescribed during treatment cycles.

CINV (chemotherapy-induced nausea and vomiting) is the most dreaded side effect before starting chemotherapy in both genders and across all age classes, and women are significantly more concerned about it than men. Patients with gynecological cancer represent an extremely challenging population in which to treat or control CINV. Indeed, female sex is associated with a higher risk of CINV. In addition, gynecological malignancies often disseminate in the abdomen, increasing the emetogenic potential of chemotherapies. Thus, these patients are at a relatively high risk of experiencing CINV.

This is a phase IV, multicentric, single arm study using a fixed dose combination of netupitant and palonsetron NEPA in the treatment of chemo-naive patients ≥18 years of age with histologically or cytologically confirmed diagnosis of endometrial cancer who will receive a single line of taxane-platinum combination with or without immunotherapy.

This study aims also to evaluate patients' expectation and perception of CINV and other chemotherapy side effects (CSEs); impact of CINV and others CSEs on quality of life, health, family and personal relationships, daily activities and employment in patients with endometrial cancer receiving paclitaxel and carboplatin regimen. The agreement between patients' assessment of CINV and other CSEs as reported in a self-report scale and what they referred to clinicians about nausea and CSEs at the following chemotherapy cycle and agreement between patients' expectation of CINV and other CSEs before initiating of chemotherapy and the side effects that they actually experienced during chemotherapy will be also evaluated.

Patients will be observed over a duration of 4 cycles. The primary endpoint will be assessed at cycle 1.

This study will enroll female patients ≥18 years of age with histologically or cytologically confirmed diagnosis of endometrial cancer who will receive a single line of taxane-platinum combination therapy with or without immunotherapy. This includes chemotherapy naïve patients who will receive taxane-platinum combination therapy in adjuvant setting or chemotherapy naïve patients who will receive first line taxane-platinum combination therapy with or without immunotherapy for primary advanced or recurrent disease. The planned number of patients is 84, and 8 centers will be involved in the trial.

Primary objective: To evaluate effectiveness of a single oral dose of NEPA in terms of complete response (CR: no emesis, no rescue medication) in the overall phase (0-120h) at cycle 1 in chemotherapy-naïve patients with endometrial cancer receiving paclitaxel and carboplatin with or without immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Subject is at least 18 years of age, able to understand the study procedures, and agrees to participate in the study by providing written informed consent
* Subject has histologically or cytologically proven endometrial cancer
* Patients were required to have an Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2
* Adequate organ function allowing the patient to receive taxane-platinum combination therapy with or without immunotherapy according to clinical practice and opinion of treating physician
* Naive to chemotherapy
* Women of child-bearing potential must have a negative pregnancy test (urine). Female patients are considered of child-bearing potential following menarche and until becoming post-menopausal unless permanently sterile. Permanent sterilization methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy. Patients are considered to not be of child-bearing potential if they have a history of tubal ligation or hysterectomy or are post-menopausal with a minimum of 1 year without menses. Patients of child-bearing potential must agree to adequate birth control if conception is possible during the study and for 6 months after the last dose; in this case, patients must take a monthly pregnancy test for the duration of the study

Exclusion Criteria:

* They will experience emesis within the 24 hours before receipt of 1 course of chemotherapy
* will be scheduled to radiation therapy to the abdomen or pelvis within 1 week before day 1 or between day 1 and 5
* Will be scheduled to undergo bone marrow or stem-cell transplant
* Chronic systemic corticosteroid use
* Brain metastasis
* Subject is considered a poor medical risk due to a serious, uncontrolled medical disorder
* History or predisposition to cardiac conduction abnormalities, torsade des pointes or severe cardiovascular diseases
* Subject is pregnant or breastfeeding or is expecting to conceive children within the projected duration of the study, starting with the screening visit through 180 days after the last dose of study treatment
* They have any known hypersensitivity or contraindication to the components of the study drugs (hypersensitivity to the active substance or to any of the excipients contained in the product, as listed in the relevant section of the summary of product characteristics)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — This study will enroll female patients ≥18 years of age with histologically or cytologically confirmed diagnosis of endometrial cancer
Enrollment: 84 (Estimated)
Dates: Start 2024-02-26 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Effectiveness | overall phase (0-120 hours after NEPA administration) at cycle 1
  Evaluate effectiveness of a single oral dose of NEPA in terms of complete response (CR: no emesis, no rescue medication) in the overall phase (0-120h) at cycle 1 in chemotherapy-naïve patients with endometrial cancer receiving paclitaxel and carboplatin chemotherapy with or without immunotherapy

SECONDARY OUTCOMES:
Effectiveness | acute (0-24 hours), delayed (>24 to 120 hours), and overall (0-120 hours) phases after the start of chemotherapy of each cycle
  Effectiveness of a single oral dose of NEPA in terms of CR and complete control (CC: no rescue medication, no emesis and no nausea (VAS score of <25 mm) during the acute (0-24 hours), delayed (>24 to 120 hours), and overall (0-120 hours) phases after the start of chemotherapy of each cycle
Effectiveness | acute (0-24 hours), delayed (>24 to 120 hours), and overall (0-120 hours) after the start of chemotherapy of each cycle
  Effectiveness of a single dose of NEPA in terms of no rescue medication, no emesis and no significant nausea (VAS score of <25 mm) during the acute (0-24 hours), delayed (>24 to 120 hours), and overall (0-120 hours) after the start of chemotherapy of each cycle
Effectiveness | acute (0-24 hours), delayed (>24 to 120 hours), and overall (0-120 hours) phases after the start of each cycle
  Effectiveness of a single oral dose of NEPA in terms of CR and complete control during the acute (0-24 hours), delayed (>24 to 120 hours), and overall (0-120 hours) phases after the start of each cycle according to Patient Emetogenicity Risk Profile assessed with CINV Risk Assessment tool
Safety | From cycle 1 to cycle 4 of the treatment
  Evaluate safety of NEPA when given in multiple treatment cycles in patients with endometrial cancer receiving paclitaxel and carboplatin regimen with or without immunotherapy
Quality of Life | during each cycle of treatment
  Evaluate QoL of patients with endometrial cancer treated with paclitaxel and carboplatin regimen receiving NEPA as antiemetic treatment in terms of FLIE scores during each cycle.
  This study aims also to evaluate patients' expectation and perception of CINV and other chemotherapy side effects (CSEs); impact of CINV and others CSEs on quality of life, health, family and personal relationships, daily activities and employment in patients with endometrial cancer receiving paclitaxel and carboplatin regimen. The agreement between patients' assessment of CINV and other CSEs as reported in a self-report scale and what they referred to clinicians about nausea and CSEs at the following chemotherapy cycle and agreement between patients' expectation of CINV and other CSEs before initiating of chemotherapy and the side effects that they actually experienced during chemotherapy will be also evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Monika Ducceschi, MD, Principal Investigator — Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Locations (8):
- Italy (8):
  - ASST Spedali Civili di Brescia, Brescia, BS
  - ASST Lecco - A. Manzoni Hospital, Lecco, LC
  - Istituto Oncologico Veneto, Padua, PD
  - Centro di Riferimento Oncologico (CRO) IRCCS, Aviano, PN
  - Azienda Ospedaliera Ordine Mauriziano di Torino, Torino, TO
  - AOU Città della Salute e della Scienza di Torino, Torino, TO
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - Istituto Europeo di Oncologia, Milan